CLINICAL TRIAL: NCT02533037
Title: Effects Of Rehabilitation Incorporating Gait Training On Clinical Measures Associated With Chronic Ankle Instability
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Jay Hertel, PhD, ATC, Professor, Department of Kinesiology, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16992
Record Dates: First submitted 2015-08-21; First posted 2015-08-26 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Chronic Ankle Instability

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Traditional Instability Tools (Active Comparator): Participants will use traditional instability tools during the impairment-based rehabilitation intervention.
  Interventions: Other: Traditional Instability Tools
- Ankle destabilization shoes (Experimental): Participants will use ankle destabilization shoes during the impairment-based rehabilitation intervention.
  Interventions: Other: Ankle Destabilization Shoes

INTERVENTIONS:
Other: Traditional Instability Tools — Participants will complete 12 sessions over 4-weeks of impairment-based rehabilitation that incorporates ankle range of motion, ankle strength, balance, and functional activity exercises. For the balance and functional activity exercises, participants will use traditional instability tools.
  Arms: Traditional Instability Tools
Other: Ankle Destabilization Shoes — Participants will complete 12 sessions over 4-weeks of impairment-based rehabilitation that incorporates ankle range of motion, ankle strength, balance, and functional activity exercises. For the balance and functional activity exercises, participants will use ankle destabilization shoes.
  Arms: Ankle destabilization shoes

SUMMARY:
This is a randomized controlled trial (RCT) regarding the conservative treatment of chronic ankle instability (CAI) with an impairment based rehabilitation program. Individuals with CAI have deficits in neuromuscular control and altered gait patterns. Ankle destabilization shoes are used clinically and may improve neuromuscular control by increasing lower extremity muscle activation, which may improve gait patterns. The investigators' purpose is to determine whether a 4-week rehabilitation program that includes ankle destabilization shoes (experimental) has beneficial effects on self-reported function and ankle gait kinematics compared to traditional rehabilitation without destabilization shoes (control) in CAI patients. In addition, the investigators will compare ankle strength and balance between CAI patients and healthy individuals with no history of ankle injury prior to the 4-week rehabilitation. The investigators hypothesize the experimental group will have greater improvement in self-reported function and frontal and sagittal plane kinematics during walking compared to the control group. In addition, the investigators hypothesize that patients with CAI will have a decrease in ankle strength and balance when compared to healthy individuals. The design is a single-blinded randomized controlled trial. Forty CAI patients will complete baseline self-reported function questionnaires and walking gait trials and then be randomized into control and experimental groups. Both groups will complete 4-weeks of supervised rehabilitation with or without destabilization shoes and then repeat the questionnaires and walking trials.

ELIGIBILITY:
Inclusion Criteria:

* CAI with a history of recurrent ankle sprains, with the first sprain occurring longer than 12 months ago. Participants will have lingering symptoms, and disability, but have not actively sought treatment for their CAI
* All participants will be physically active: Participating in some form of physical activity for at least 20 min per day, three times per week.

Exclusion Criteria:

* Neurological or vestibular disorders affecting balance
* Currently seeking medical care for CAI
* History of prior ankle surgery
* History of ankle sprain within the past 6 weeks
* History of ankle fracture
* Diabetes mellitus
* Current self-reported disability due to lower extremity pathology that may adversely affect neuromuscular function
* Lumbosacral radiculopathy
* Pregnant
* Soft tissue disorders including Marfan's syndrome and Ehlers-Dandros syndrome

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2013-08; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in self-reported function as measured by the Foot and Ankle Ability Measure questionnaire | after 4-weeks of rehabilitation
  Scores range from 100%(no decrease in function) to 0%(complete loss of function)

SECONDARY OUTCOMES:
Changes from baseline in ankle range of motion measured in degrees | after 4-weeks of rehabilitation
  Four different ankle ranges of motion will be measured using a bubble inclinometer
Changes from baseline in ankle maximum voluntary isometric strength | after 4-weeks of rehabilitation
  Ankle maximum voluntary isometric strength will be measured during five different ankle positions using a hand-held dynamometer.
Changes from baseline in balance | after 4-weeks of rehabilitation
  Static balance will be measured by participants standing on one limb on a forceplate to measure the participant's center of pressure.
Changes from baseline in lower extremity electromyography during ankle maximal voluntary isometric strength testing | after 4-weeks of rehabilitation
  Lower extremity electormyography during maximal isometric strength testing will be measured using surface EMG electrodes over the peroneus brevis, peroneus longus, anterior tibialis, and medial gastrocnemius muscles.
Changes from baseline in lower extremity electromyography during balance | after 4-weeks of rehabilitation
  Lower extremity electormyography during balance testing will be measured using surface EMG electrodes over the peroneus brevis, peroneus longus, anterior tibialis, and medial gastrocnemius muscles.
Changes from baseline in lower extremity kinematics during walking | after 4-weeks of rehabilitation
  Ankle, knee, and hip motion during walking measured by a 3D motion capture system
Changes from baseline in lower extremity kinetics during walking | after 4-weeks of rehabilitation
  Ankle, knee, and hip moments during walking measured by a 3D motion capture system
Changes from baseline in lower extremity surface electromyography during walking | after 4-weeks of rehabilitation
  Lower extremity electormyography during walking will be measured using surface EMG electrodes over the peroneus brevis, peroneus longus, anterior tibialis, and medial gastrocnemius muscles.

CONTACTS AND LOCATIONS:
Overall Officials: Jay Hertel, PhD, ATC, Principal Investigator — University of Virginia